CLINICAL TRIAL: NCT06690099
Title: Prospective Collection of Whole Blood Specimens From RhD Negative Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: Devyser Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DVYUS-RHD-001
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Rhesus D Genotype; Pregnancy
Keywords: RhD negative; fetal DNA; cell free fetal DNA; Fetal RhD genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human blood specimens will be processed to plasma and stored for future use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who are RhD negative and between 12 and 28 weeks gestation

SUMMARY:
The purpose of this research is to collect blood samples and data from pregnant women who are Rh negative. The blood will be used for the future research and the development of non-invasive prenatal tests to identify Rh blood type status of the baby during pregnancy.

DETAILED DESCRIPTION:
This is a prospective multi-center blood collection study. Women 18 years of age or older with a viable singleton pregnancy between12 weeks and 28 weeks gestation will be enrolled.

Whole blood samples will be collected from each enrolled patient. Maternal specimens will be processed to plasma and stored for future testing with non-invasive prenatal tests to identify fetal Rh status.

Baby RhD blood type status will be recorded after delivery. All obstetric clinical management will take place per standard clinic practices and procedures and will not be altered by participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. 18 years of age or older at enrollment
3. Women with a viable pregnancy (with documented fetal heartbeat) between 12 weeks, 0 days and 28 weeks, 0 days gestational age
4. Women with RhD negative antigen status by serology
5. Willing to provide neonatal ABO and RhD genotyping status

Exclusion Criteria:

1. Women with multiple gestation pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are RhD negative and between 12 and 28 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fetal RhD determination from maternal whole blood | 18 months
  Collected samples will be used for future development of non-invasive prenatal test to determine fetal RhD status from maternal whole blood

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers. Any shared data will be de-identified data at the cohort level in aggregate.